CLINICAL TRIAL: NCT04921826
Title: Potential Causes of Retained Items During Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Imam Mohammad ibn Saud Islamic University (Other)
Responsible Party: Principal Investigator, mohammad bukhetan alharbi, associate professor, Imam Mohammad ibn Saud Islamic University
Other Study IDs: RETAINED ITEM DURING SURGERY
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Foreign Bodies; Surgical Sponge, Retained
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: online survey — online survey

SUMMARY:
to understand and analyze the potential causes of retained items (sponge and instruments) during surgery, which include room preparations, initial count, adding sponges, removing sponges, first closing count, final closing count.

ELIGIBILITY:
Inclusion Criteria:

• operating room staff of hail hospital cluster

Exclusion Criteria:

• none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: an online survey will be send through cluster administration to operating room staff ,to answer voluntarily without compensation. informed consent was obtained. This study was exempt from review board approval at authors' institutions.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
study potential causes of retained item during surgery | 20 days
  to understand participant opinion about the potential causes of retained item which include :room preparation with needed operating room equipment according to the specialty, initial count of sponges and instruments, adding sponges by event recording in a chart, removing sponges by event recording in a chart, first closing count in a chart , final closing count in a chart.

CONTACTS AND LOCATIONS:
Overall Officials: mohammad alharbi, Principal Investigator — imam mohamamd ibn saud islamic university
Locations (1):
- Hail Health Cluster, Hail, Other, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided